CLINICAL TRIAL: NCT05584852
Title: Prognostic Value of Myosteatosis and Creatinine-to-cystatin C Ratio in Patients With Resectable Pancreatic Ductal Adenocarcinoma
Brief Title: Prognostic Value of Myosteatosis and Creatinine-to-cystatin C Ratio in Patients With Pancreatic Ductal Adenocarcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Principal Investigator, jingxue, Prof, The Affiliated Hospital of Qingdao University
Other Study IDs: QYFYWZLL27348
Record Dates: First submitted 2022-10-14; First posted 2022-10-18 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Skeletal Muscle Radiodensity; Myosteatosis; Scr/CysC Ratio; Pancreatic Ductal Adenocarcinoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- with myosteatosis
- without myosteatosis

INTERVENTIONS:
Other:  — no intervention

SUMMARY:
Pancreatic ductal adenocarcinoma (PDAC) is a dismal disease with a 5-year survival rate as low as 6%. It causes body composition changes and many patients develop muscle loss with disease progression. Computed tomography (CT) is a common, noninvasive method of muscle assessment.Known as myoesteatosis,low muscle radiodensity is reflective of intermuscular adipose tissue that influences survival outcomes in patients with cancer.Serum creatinine (Scr) and cystatin C (CysC) are usually employed to estimate renal function in clinical practice. Scr is a metabolic waste product produced by creatine in skeletal muscle. CysC can be produced by all nucleated cells in the body at a constant production rate. CysC is used as an endogenous marker to reflect the glomerular filtration rate. Some studies have supported that the Scr/CysC ratio (CCR) is a simple and inexpensive measure that can be used to evaluate the skeletal muscle mass of patients with malignancies, such as gastric cancer. Therefore, the purpose of the present study is to explore the association between CCR and myosteatosis upon diagnosis of PDAC, specially whether the co-occurrence of these factors could predict survival outcomes.Preoperative assessment of muscle quality may be valuable for treatment planning and optimization of nutritional support.

This retrospective study enrolls patients who underwent surgery for PDAC, from January 2016 to December 2021. Patients will be divided into myosteatosis and non-myosteatosis groups. Clinical and imaging data are collected.The study does not have any intervention measures and harm to subjects.

DETAILED DESCRIPTION:
Inclusion criteria:

a）aged between 18 and 75; b) pancreatic ductal adenocarcinoma confirmed by biopsy or postoperative pathology; c) CT and renal function related data within 1 month before operation; d) voluntarily participate in this study and have informed consent.

Exclusion criteria:

* pancreatic malignant tumors of other pathological types or other malignant tumors;

  * received local or systemic radiotherapy and chemotherapy before operation; ③ with severe metabolic diseases such as decompensated cirrhosis, nervous system diseases and muscle degenerative diseases; ④ absent of preoperative imaging or clinical data;

ELIGIBILITY:
Inclusion Criteria:

* a） aged between 18 and 75; b) pancreatic ductal adenocarcinoma confirmed by biopsy or postoperative pathology; c) CT and renal function related data within 1 month before operation; d) voluntarily participate in this study and have informed consent.

Exclusion Criteria:

* ① pancreatic malignant tumors of other pathological types or other malignant tumors;

  * received local or systemic radiotherapy and chemotherapy before operation;

    * with severe metabolic diseases such as decompensated cirrhosis, nervous system diseases and muscle degenerative diseases; ④ absent of preoperative imaging or clinical data; ⑤ Lost interviewers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective study enrolled patients who underwent surgery for resectable pancreatic ductal adenocarcinoma, from January 2016 to December 2021. Patients will be divided into myosteatosis and non-myosteatosis groups according to skeletal muscle radiodensity.
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
overall survival | 2016.1.1-2022.12.31
  Time from operation to death or the last follow-up
Disease free survival | 2016.1.1-2022.12.31
  Time from operation to recurrence or the last follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- the Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No